CLINICAL TRIAL: NCT05151510
Title: A Randomized Controlled Study Comparing Trigger Point Injections With 1% Lidocaine Versus 5% Lidocaine Patch for Myofascial Pain in the Emergency Department
Brief Title: Trigger Point Injections Versus Lidocaine Patch for Myofascial Pain in the Emergency Department
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCI IRB HS# 2021-6439
Record Dates: First submitted 2021-09-08; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Myofascial Trigger Point Pain; Myofacial Pain
Keywords: pain management; emergency department; trigger point injections; lidocaine patches; myofascial pain; interventional pain medicine
MeSH Terms: conditions — Myofascial Pain Syndromes; Facial Pain; Agnosia; Emergencies | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This will be a single-center, prospective, randomized, pragmatic trial carried out with patients that have a primary complaint of myofascial back and/or posterior neck pain. Upon presentation to the emergency department, if the patient is found to have myofascial pain, they will be approached by research personnel to be enrolled in the study. If the patient consents to be in the study, the patient will then be randomly assigned to either receive a trigger point injection or receive lidocaine patch (5%) therapy. The lidocaine patch therapy group cannot receive a trigger point injection. Randomization will occur in blocks of 2, using a Web- based randomization program (http://sealedenvelope.com).
Who Masked: Outcomes Assessor
Masking Description: Given the trigger point injection is physician performed, and very different from placing a lidocaine patch, we cannot blind investigators nor the patient to the intervention. We will, however, blind our outcome assessors in regards to which intervention the patient had received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trigger point with 1% Lidocaine (Experimental): The physician will withdraw 1cc of 1% lidocaine in a 25g needle, sterilely prep the field with a Chloraprep applicator, use index, and middle finger to squeeze the borders of the trigger point and raise the central aspect of the trigger point, insert the needle at 90-degree angle up to 5/8' deep, inject 1cc of the 1% lidocaine after ensuring needle is not in a blood vessel, removing the needle, and then covering the insertion site with a sterile bandage.
  Interventions: Procedure: Trigger point injection with 1% lidocaine
- 5% Lidocaine Patch (Active Comparator): 5% lidocaine patch will be placed at the point of maximal tenderness upon palpation. Location of placement will be described and instructed by physician and placed by nursing staff.
  Interventions: Drug: Lidocaine patch 5%

INTERVENTIONS:
Procedure: Trigger point injection with 1% lidocaine — Previously discussed in prior section.
  Arms: Trigger point with 1% Lidocaine
Drug: Lidocaine patch 5% — Will place lidocaine patch onto skin overlaying point of maximal tenderness
  Arms: 5% Lidocaine Patch

SUMMARY:
The aim of this trial is to investigate the efficacy of trigger point injections with 1% lidocaine in reducing myofascial back and neck pain in the Emergency Department compared to lidocaine patches 5%.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks and benefits, all patients will be randomized into either the trigger point injection group with 1% lidocaine, or the 5% lidocaine patch group. Pain scores will be recorded while in the emergency department, and we will have a 5 day follow-up phone call to assess efficacy. Patients who present to UCI Department of Emergency medicine will be screened and recruited prospectively, and information regarding this study will be available on clinicaltrials.gov as a method of recruitment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with myofascial pain of the posterior neck or back. *The diagnosis of myofascial pain was based on established criteria of having a palpable taut band (trigger point) that when depressed reproduced the patient's pain.

Exclusion Criteria:

* midline spinal tenderness
* evidence of radiculopathy
* pregnant
* have an allergy to lidocaine
* altered or deemed incapable of making informed consent
* had signs of infection or skin breakdown over the trigger point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
absolute change in Numerical Rating Scale (NRS) of pain | 0 minutes and 20-minutes post- treatment, and every 30-60 minutes thereafter until discharge or admission and we will give the patient a hand out so that they can record their pain scores for up to 5 days after their emergency department visit.
  Pain on a scale of 1-10. Minimum value is 1, maximum value is 10. Higher score means higher level of pain while lower score means lower level of pain.

SECONDARY OUTCOMES:
use of other medications for treatment of pain including medications administered | From initiation of the study up to 5 days post discharge
  How often and which medications did the patient require in emergency department and upon discharge to control their pain
disposition times | From initiation of the study up to the point the patient is discharged from the emergency department
  Number of minutes it takes to discharge or admit the patient from first contact
satisfaction/experience surveys regarding their treatment | Immediately after the intervention is performed/administered
  We will administer satisfaction/experience surveys to assess for any discomfort or relief from the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lee, MD, Principal Investigator — UCI Department of Emergency Medicine
Locations (1):
- Emergency Room at UCI Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yanuck J, Saadat S, Lee JB, Jen M, Chakravarthy B. Pragmatic Randomized Controlled Pilot Trial on Trigger Point Injections With 1% Lidocaine Versus Conventional Approaches for Myofascial Pain in the Emergency Department. J Emerg Med. 2020 Sep;59(3):364-370. doi: 10.1016/j.jemermed.2020.06.015. Epub 2020 Jul 22. PMID 32712034
- [Background] Skootsky SA, Jaeger B, Oye RK. Prevalence of myofascial pain in general internal medicine practice. West J Med. 1989 Aug;151(2):157-60. PMID 2788962
- [Background] Scott NA, Guo B, Barton PM, Gerwin RD. Trigger point injections for chronic non-malignant musculoskeletal pain: a systematic review. Pain Med. 2009 Jan;10(1):54-69. doi: 10.1111/j.1526-4637.2008.00526.x. Epub 2008 Nov 5. PMID 18992040
- [Background] Garvey TA, Marks MR, Wiesel SW. A prospective, randomized, double-blind evaluation of trigger-point injection therapy for low-back pain. Spine (Phila Pa 1976). 1989 Sep;14(9):962-4. doi: 10.1097/00007632-198909000-00008. PMID 2528826
- [Background] Annaswamy TM, De Luigi AJ, O'Neill BJ, Keole N, Berbrayer D. Emerging concepts in the treatment of myofascial pain: a review of medications, modalities, and needle-based interventions. PM R. 2011 Oct;3(10):940-61. doi: 10.1016/j.pmrj.2011.06.013. PMID 22024326
- [Background] Affaitati G, Fabrizio A, Savini A, Lerza R, Tafuri E, Costantini R, Lapenna D, Giamberardino MA. A randomized, controlled study comparing a lidocaine patch, a placebo patch, and anesthetic injection for treatment of trigger points in patients with myofascial pain syndrome: evaluation of pain and somatic pain thresholds. Clin Ther. 2009 Apr;31(4):705-20. doi: 10.1016/j.clinthera.2009.04.006. PMID 19446144